CLINICAL TRIAL: NCT04532567
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of GLPG1205 for 14 Days in Healthy Japanese and Caucasian Male Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GLPG1205 in Healthy Japanese and Caucasian Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG1205-CL-121
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GLPG1205 dose A (Experimental): Participants will receive a single dose with dose A of GLPG1205 on Day 1 in Period 1, and 14 days q.d. dosing on Days 1 to 14 in Period 2.
  Interventions: Drug: GLPG1205
- Placebo dose A (Placebo Comparator): Participants will receive a single dose placebo on Day 1 in Period 1, and 14 days q.d. dosing on Days 1 to 14 in Period 2.
  Interventions: Drug: Placebo
- GLPG1205 dose B (Experimental): Participants will receive 14 days q.d. dosing with dose B of GLPG1205 on Days 1 to 14.
  Interventions: Drug: GLPG1205
- Placebo dose B (Placebo Comparator): Participants will receive 14 days q.d. dosing placebo on Days 1 to 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1205 — GLPG1205 film-coated tablets
  Arms: GLPG1205 dose A; GLPG1205 dose B
Drug: Placebo — placebo film-coated tablets
  Arms: Placebo dose A; Placebo dose B

SUMMARY:
The purpose of this research study is to assess the safety and tolerability of GLPG1205 in single and multiple oral doses in healthy male Caucasian and Japanese subjects. This study will also assess the pharmacokinetics (PK) across different doses of GLPG1205. PK will look at how the study drug is absorbed, broken down, and eliminated by your body.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian and Japanese male between 20-55 years of age (extremes included), on the date of signing the informed consent form (ICF).
* Japanese subjects must be first generation Japanese of full Japanese parentage, and must have not lived outside Japan for more than 5 years. First generation subjects will have been born in Japan of 2 parents and 4 grandparents also born in Japan of full Japanese descent.
* A body mass index (BMI) between 18-26 kg/m2, extremes included, with a minimum body weight of 45 kg.
* Able and willing to comply with the protocol requirements and signing the ICF as approved by the Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to any screening evaluations.

Exclusion Criteria:

* History of serious allergic reaction to any drug as determined by the investigator (e.g., anaphylaxis requiring hospitalization) and/or known sensitivity to the investigational product (IP) or its excipients as determined by the investigator.
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first dosing of the IP.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuation | From screening through study completion, an average of 3 months
  To evaluate the safety and tolerability of single and multiple oral doses of GLPG1205 in healthy male Japanese and Caucasian subjects
Maximum observed plasma concentration (Cmax) of GLPG1205 | Between Day 1 pre-dose and Day 18 and at follow-up Day 32
  To assess the PK of single and multiple oral doses of GLPG1205 in healthy male Japanese subjects matched with healthy male Caucasian subjects
Area under the plasma concentration-time curve from time zero till 24 hours postdose (AUC 0-24h) of GLPG1205 | Between Day 1 pre-dose and Day 18 and at follow-up Day 32
  To assess the PK of single oral doses of GLPG1205 in healthy male Japanese subjects matched with healthy male Caucasian subjects
Area under the plasma concentration-time curve over the dosing interval (AUC T) of GLPG1205 | Between Day 1 pre-dose and Day 18 and at follow-up Day 32
  To assess the PK of multiple oral doses of GLPG1205 in healthy male Japanese subjects matched with healthy male Caucasian subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Tankisheva, MD, PhD, Study Director — Galapagos NV
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No